## STATISTICAL ANALYSIS PLAN

STUDY NUMBER: SLI-C40-001
Study Part A (Excisions)

Version: v. 1.0

Date: 09-Oct-2020

Safety and Efficacy of SLI-F06 in Wound Healing and Scar Appearance in Pre-Abdominoplasty Surgical Excisions and Post-Operative Scar Appearance in Subjects Undergoing Abdominoplasty

## **Study Sponsor**

Scarless Laboratories Inc. 369 South Doheny Drive, Suite 1201 Beverly Hills, CA USA 90211

## **Clinical Research Organization**

ethica CRO Inc. 8555 Transcanada Hwy, Suite 201 Montreal, Canada H4S 1Z6 866-384-4221

#### **Confidentiality Statement**

The information contained in this document is provided in confidence. It is understood that this information will not be disclosed to others without prior agreement with the Sponsor, except to other study personnel and to the extent necessary to obtain informed consent from participating subject.

v.1.0; 09-Oct-2020 

# SAP APPROVAL SIGNATURE PAGE

The following individuals approve this version of the SLI-C40-001 Part A Statistical Analysis Plan.

| Accepted for the Sponsor – Scarless Laboratories Inc. | |
|---|---|
| Daine 1 No. | |
| Printed Name | Title |
| Signature | Date |
| Accepted for the Clinical | Research Organization - ethica CRO Inc. |
| Printed Name | Title |
| Signature | Date |

v.1.0; 09-Oct-2020 

# TABLE OF CONTENTS

| SAP | APPRO | VAL SIGNATURE PAGE | 2 |
|-----|-----------------|----------------------------------------|----|
| ГАВ | LE OF | CONTENTS | 3 |
| ABB | REVIA | ΓΙΟΝS | 4 |
| 1 | INT | RODUCTION | 5 |
| | 1.1 | Background | |
| | 1.2 | Objectives | |
| | 1.3 | Study Design | |
| 2 | STU | DY POPULATION | |
| 3 | TRE | ATMENT ALLOCATION AND RANDOMIZATION | 8 |
| 4 | STU | DY EVALUATIONS | 8 |
| | 4.1 | Primary Efficacy Variable | |
| | 4.1.1 | POSAS (PI Assessment) – Excisions | 8 |
| | 4.2 | Secondary Efficacy Variables | 8 |
| | 4.2.1 | Histology | 8 |
| | 4.2.2 | Tensile Strength | 8 |
| | 4.3 | Exploratory Efficacy Variable | 8 |
| | 4.3.1 | POSAS (Subject Assessment) – Excisions | 8 |
| | 4.4 | Safety Variables | 8 |
| | 4.4.1 | Adverse Events (AEs) | 8 |
| | 4.4.2 | Clinical Safety Laboratory Tests | 8 |
| | 4.4.3 | Immunogenicity Testing | 8 |
| | 4.4.4 | | |
| 5 | ANA | ALYSIS POPULATIONS | 9 |
| 3 | 5.1 | Populations | |
| | 5.1.1 | 1 | |
| | 5.1.2 | , , <u>.</u> | |
| | 5.1.3 | | |
| _ | | | |
| 6 | | IPLE SIZE JUSTIFICATION | |
| 7 | | TISTICAL METHODS | |
| | 7.1 | Efficacy Analyses | |
| | 7.2 | Safety Analyses | |
| | 7.3 | Adverse Events (AEs) | |
| | 7.4 | Concomitant Medications and Procedures | |
| | 7.5 | Safety Laboratory Tests | |
| | 7.6 | Immunogenicity | |
| | 7.7 | General Statistical Considerations | |
| | 7.7.1 | | |
| | 7.7.2 | 1 | |
| | 7.7.3 | e | |
| | 7.7.4 | 1 | |
| | 7.7.5 | 1 1 | |
| | 7.7.6 | | |
| | 7.7.7 | | |
| | 7.7.8 | Outliers | 11 |
| | <b>Δ DDENII</b> | DIX A: SUMMARY OF STATISTICAL TESTS | 12 |
| | | DIX A. SUMMART OF STATISTICAL TESTS | 14 |

# **ABBREVIATIONS**

| AE | Adverse Event |
|---------------|-------------------------------------------------|
| BL | Baseline |
| BMI | |
| | Body Mass Index |
| CFR | U. S. Code of Federal Regulations |
| CTR | Common Treatment Response |
| CRO | Clinical Research Organization |
| DP | Drug Product |
| Excision site | A mapped area designated for a single excision. |
| eCRF | electronic Case Report Form |
| IRB | Institutional Review Board |
| ITT | Intent-to-Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PI | Principal Investigator |
| POC | Proof Of Concept |
| POSAS | Patient and Observer Scar Assessment Scale |
| PP | Per protocol |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAFT | Safety |
| SAP | Statistical Analysis Plan |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| TRAE | Treatment Related Adverse Event |
| Tx | Treatment |
| UPT | Urine Pregnancy Test |
| USP | United States Pharmacopeia |

v.1.0; 09-Oct-2020 

#### 1 INTRODUCTION

This statistical analysis plan (SAP) gives a comprehensive and detailed description of statistical techniques to be used for study SLI-C40-001. The purpose of this SAP is to ensure the credibility of the study findings by pre-specifying the statistical approaches for the analysis of study data prior to database lock. This SAP provides additional details concerning the statistical analyses outlined in the protocol. Whenever differences exist in descriptions or explanations provided in the protocol and SAP, the SAP prevails.

#### 1.1 Background

SLI-F06 is a synthetic peptide that is being developed as a treatment to promote wound healing and improve scar appearance. The amino acid sequence of SLI-F06 is derived from an endogenous human protein that has been shown in animal models to promote accelerated wound healing, reduced scarring, and increased wound tensile strength. In these same animal models, the SLI-F06 has been demonstrated to retain similar pro-migration, pro-tensile strength, and anti-fibrotic properties as the endogenous protein.

SLI-F06 drug product (DP) is a sterile lyophilized powder consisting of SLI-F06 as the active ingredient and formulation buffer components. The DP will be reconstituted in clinic with USP Water for Injection and injected intradermally along both edges of a freshly made excision to achieve a primarily local effect.

The study population will consist of healthy patients planning to undergo elective abdominoplasty. During **Part A** of this study (i.e., Phase I Safety/Proof of Concept), each subject will receive 12, 14, or 18 small or large excisions at 8 weeks or 12 weeks pre-abdominoplasty. Wounds treated with SLI-F06 or vehicle will be followed until the time of abdominoplasty when the tissue is harvested. At the completion of study Part A, subjects will enter study **Part B** where they will undergo the abdominoplasty, have the abdominoplasty incision treated with SLI-F06, and be followed for an additional 12 months.

# This SAP covers Study Part A only

v.1.0; 09-Oct-2020 

## 1.2 Objectives

The primary objectives of this study are the following:

 Assess the safety and tolerability of SLI-F06 in the treatment of planned surgical excisions.

Secondary objectives include, but are not limited to, the following:

- Assess the effect of SLI-F06 on post-excisional scar appearance.
- Assess the effect of SLI-F06 on wound strength.
- Assess the effect of SLI-F06 on histological appearance of scars.
- Assess immunogenicity effects of SLI-F06.

## 1.3 Study Design

This is a multicenter, double-blind study comparing the safety of SLI-F06 to control formulation buffer (vehicle), as well as comparing the improvement in scar appearance and wound strength. Each subject will serve as his or her own control. The study is divided into 2 parts where Part A is a Phase I safety/proof of concept study of small scars pre-abdominoplasty, and Part B is a Phase IIa study of post-abdominoplasty scars.

In **Part A** of the study (i.e., Phase I safety/proof-of-concepts. Subjects will then be randomized by side of the pannus (right or left) for treatment with SLI-F06 or formulation buffer, wound tension (high or low), and by duration of follow-up post-excisions to 12 weeks (group 1) or 8 weeks (group 2) pre-abdominoplasty. Excision mapping and number of excisions will be determined by size of pannus as follows:

- Small pannus: 6 low tension and 6 high tension wounds will (12 wounds/subject).
- Medium pannus: 6 low tension and 8 high tension wounds will (14 wounds/subject).
- Large pannus: 8 low tension and 10 high tension wounds (18 wounds/subject).

Following completion of the follow-up period, the entire abdominoplasty site will be harvested and sent for analyses of histopathology and tensile strength.

In **Part B** of the study (i.e., Phase IIa), <u>ALL</u> subjects who complete Part A will be randomly assigned to receive injections of SLI-F06 along one half (left or right) of the abdominoplasty incision and control injections along the other half. The subject will undergo routine wound care and will attend study follow-up visits following abdominoplasty at Day 8 and at Months 1, 2, 3, 6, 9, and 12.

v.1.0; 09-Oct-2020 

Scarless Laboratories
SLI-C40-001 – SAP (Study Part A)
CONFIDENTIAL

## **STUDY SUMMARY**

| | | Part A (P | hase I Safety/P | roof of C | Concept) | | Part B (Phase IIa) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | 1a | 2a | 3a | 4a | 5a | 6a | 1b | 2b | SR | 3b | 4b | 5b | 6b | 7b | 8b |
| Assessment and Procedures | Screening<br>Period | Excisions | Suture<br>Removal | | | | Abdomin-<br>oplasty | | Suture<br>Removal | | | | | | |
| Assessment and 11 occurres | D -30<br>to 0 | D1 | D8<br>± 1d | D29<br>± 2d | D57<br>± 3d | D85<br>± 3d | D0 | D8<br>± 1d | PI<br>Discretion | M1<br>± 3d | M2<br>± 7d | M3<br>± 14d | M6<br>± 14d | M9<br>± 14d | M12<br>± 14d |
| Informed Consent | X | | | | | | | | | | | | | | |
| Inc/Excl Criteria | X | | | | | | | | | | | | | | |
| Medical/Surgical History | X | | | | | | | | | | | | | | |
| Physical Exam | X | | | | | | | | | | | | | | |
| Urine Pregnancy Test <sup>1</sup> | X | X 1 | | | | | X | | | | | X | X | X | X |
| Abdominoplasty Area Assessment & selection of Pannus Map size | X | | | | | | | | | | | | | | |
| Immunogenicity sampling | X | | X | X | X | X | | X | | X | X | X | X | X | X |
| Safety Laboratory Testing <sup>2</sup> | X 2 | | | X | Group 2 | Group 1 | | | | X | | | | | X |
| Photography <sup>3</sup> | | X 3 | X 3 | X | X | X | | | | X | X | X | X | X | X |
| Randomization | | X | | | | | X | | | | | | | | |
| Excisions | | X | | | | | | | | | | | | | |
| IP Injections | | X | | | | | X | | | | | | | | |
| Abdominoplasty/ Tissue<br>Harvesting | | | | | | | X | | | | | | | | |
| Suture removal | | | X | | | | | | X | | | | | | |
| POSAS grading | | | Post-removal of sutures | X | X | X | | | | X | X | X | X | X | X |
| AE Assessment | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Group 1; 12 week assessment | | | | | | | ] | | | | | | | | |
| Exit from Part A / Start of Part B | | | | | | X | Ì | | | | | | | | |
| Group 2; 8 week assessment <sup>4</sup> | | | | | | | • | | | | | | | | |
| Exit from Part A / Start of Part B | | | | | X | | | | | | | | | | |

<sup>1</sup> UPT if female of childbearing potential and if last UPT performed >7 days of V2a.

v.1.0; 09-Oct-2020

<sup>2</sup> Safety laboratory results to be reviewed by the PI prior to excisions in order to confirm absence of any health condition(s) that would make the subject inappropriate for study entry.

<sup>3</sup> Day 1 photography occurs prior to excisions and following closure of all excisions, and Day 8 photography occurs pre- and post-removal of sutures.

**<sup>4</sup>** Only **currently enrolled** participants who cannot be moved from group 2 to group 1 will remain in group 2

#### 2 STUDY POPULATION

Healthy adult subjects presenting for abdominoplasty surgery will be enrolled and randomized. The full description of the inclusion and exclusion criteria is found in Section 5 of the study protocol.

#### 3 TREATMENT ALLOCATION AND RANDOMIZATION

All excisions to be treated with SLI-F06 for a given subject will be on one side of the mapped area (i.e., left side or right side) and vehicle treated excisions will be on the other side of the mapped area.

#### 4 STUDY EVALUATIONS

#### 4.1 Primary Efficacy Variable

## 4.1.1 POSAS (PI Assessment) – Excisions

The Patient and Observer Scar Assessment Scale (POSAS) will be used to assess the various parameters of each excision site. At each observation time point, the <u>PI</u> will grade each scar using the "Observer Scale" of the POSAS.

## 4.2 Secondary Efficacy Variables

## 4.2.1 Histology

Histology of excision sites will be evaluated and reported separately from the analyses described in this SAP.

#### 4.2.2 Tensile Strength

Ex vivo tensile strength of excision sites will be assessed and compared.

#### 4.3 Exploratory Efficacy Variable

#### 4.3.1 POSAS (Subject Assessment) – Excisions

Subjects will grade the abdominoplasty scar using the "Patient Scale" criteria of the POSAS.

## 4.4 Safety Variables

#### 4.4.1 Adverse Events (AEs)

The Treating Investigator will assess AEs and record details of seriousness, severity, duration, and action taken with the study device, and relationship to the study device.

## 4.4.2 Clinical Safety Laboratory Tests

Standard clinical laboratory analyses (CBC/Diff, chemistry) will be conducted on blood samples collected at Screening V1a, V4a (D29), V5a (D57), V6a (D85). Clinically significant results, in the opinion of the PI, will be reported as AEs.

#### 4.4.3 Immunogenicity Testing

Immunogenicity analyses will be conducted on blood samples collected from subjects at Screening V1a, V3a (D8), V4a (D29), V5a (D57) and V6a (D85).

#### 4.4.4 Concomitant Medications and Procedures

Any medication or procedure (including OTC preparations) that the subject takes during the study protocol period will be considered concomitant medication and will recorded.

v.1.0; 09-Oct-2020 

#### 5 ANALYSIS POPULATIONS

## 5.1 Populations

## 5.1.1 Intent-to-Treat (ITT) Population

The ITT population will be the primary population for efficacy and safety analyses and will consist of all randomized subjects who received at least one injection of IP and provided at least one post-baseline evaluation, and will be analyzed in the treatment group they were allocated.

#### 5.1.2 Per Protocol (PP) Population

A per-protocol (PP) population will neither be identified nor analyzed.

## 5.1.3 Safety (SAFT) Population

The SAFT population will be used for safety analysis and will consist of all randomized subjects who received one injection of IP, and will be analyzed as per the treatment actually received.

#### **6** SAMPLE SIZE JUSTIFICATION

This is a Phase I safety/proof-of-concept study and a formal sample size justification is not required. It is the opinion of the Sponsor that a total of 25 subjects will be sufficient to achieve the objectives of the study.

## 7 STATISTICAL METHODS

## 7.1 Efficacy Analyses

Efficacy analyses will be conducted on an intent-to-treat (ITT) basis.

For categorical parameters, the number and percentage of subjects/observations in each category will be presented. The denominator will be based on the number of subjects/observations appropriate for the purpose of analysis. For continuous parameters, descriptive statistics will include n (number of subjects or observations), mean, standard deviation, median, and range.

Comparisons between treatment groups will be based on 95% confidence intervals.

## 7.2 Safety Analyses

Safety analysis will be conducted on the Safety Population (SAFT), by tabulations of AEs, safety laboratory parameters and immunogenicity outcomes.

## 7.3 Adverse Events (AEs)

Safety outcomes will be incidence rate of AEs, including SAEs, types of AEs and relationship to study treatment (i.e., Treatment-Emergent Adverse Events [TEAEs]; Treatment-Related-Adverse Events [TRAEs]). TEAEs will include all reported AE since the time of informed consent. TRAEs will include all reported AEs that were deemed by the Investigator to be related or not-related to study treatment.

Safety data will be tabulated with descriptive group statistics (mean, standard deviation, minimum, maximum). Severity and relationship to study treatment will be assessed.

AEs will be coded using MedDRA. These events, irrespective of relationship to study medication, will be summarized by treatment groups, MedDRA system organ class (SOC) and MedDRA preferred term (PT). The number of subjects reporting an AE, the number of AEs, and percentages of subjects in each category will be summarized. AEs by severity and relationship to study will be summarized in a similar way. Serious AEs will be summarized separately. Specifically, the following AE incidence tables will be provided:

v.1.0; 09-Oct-2020 

- Treatment-Emergent AEs: Sorted By SOC and PT
- Treatment-Related AEs: Sorted By SOC and PT
- Treatment-Emergent SAEs: Sorted By SOC and PT
- Treatment-Related SAEs: Sorted By SOC and PT

AE incidence rates with exact 95% confidence intervals will be calculated for each safety variable; confidence intervals will be used to confirm whether distribution of subjects with events is homogeneous between the treatment groups.

#### 7.4 Concomitant Medications and Procedures

Descriptive statistics (i.e., frequency and percent) will be calculated for each treatment group.

## 7.5 Safety Laboratory Tests

Determination of clinical significance for all out-of-range laboratory values will be made by each PI, and Adverse Event reports will be generated as necessary.

#### 7.6 Immunogenicity

Changes from baseline in immunogenicity outcomes will be summarized with descriptive statistics and text, as appropriate.

#### 7.7 General Statistical Considerations

#### 7.7.1 Statistical Testing

For specific information regarding the statistical tests to be used in this study, please refer to Appendix A: Summary of Statistical Tests. Comparisons between treatment groups will be based on 95% confidence intervals.

#### 7.7.2 Descriptive Statistics

Descriptive statistics (i.e., frequency and percent) will be calculated for each treatment group. Quantitative variables will be presented by way of number of observations, number of missing values, mean, standard deviation, extreme values (minimum and maximum), median, and 95% confidence internals. Categorical data will be presented by way of number of observations, number of missing values, and for each observed category, the number of occurrences and its corresponding percentage, and 95% confidence internals.

#### 7.7.3 Missing Values

Missing data will not be imputed. Data will be analyzed as observed.

#### 7.7.4 Discontinuation and Drop-Outs

Dropouts will not be replaced. All available data from dropouts will be included in the ITT analysis.

#### 7.7.5 Multiple Comparisons

No methods will be used to accommodate multiplicity (unless otherwise specified).

## 7.7.6 Multicenter Data

The data will be pooled across centers for analysis. Additionally, data for each center will be provided in data listings.

#### 7.7.7 Subject Disposition

A tabulation of subject disposition will be provided which will include the numbers of subjects

v.1.0; 09-Oct-2020 

who enter, complete, and discontinue the study. The reasons for discontinuation will be included.

## 7.7.8 Outliers

No method to process outliers will be used. Data will be analyzed as reported in the database.

v.1.0; 09-Oct-2020 

# APPENDIX A: SUMMARY OF STATISTICAL TESTS

## STUDY DISPOSITION

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Populations | Statistical<br>Tests |
|---|---|---|---|---|
| Subject discontinuations | Listing: - Last Visit - Reason for discontinuing | Exit Form | IIT | |
| Primary Reason for discontinuations | Categorical | Exit Form | IIT | |
| Disposition at each Visit | Frequency of subjects attending visit | All Visits | IIT | |
| Study dates | <ul><li>FPFV</li><li>LPFV</li><li>LPLV</li><li>Enrolment duration</li><li>Study duration</li></ul> | All Visits | IIT | |

## **BASELINE CHARACTERISTICS**

## **Demographics**

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Populations | Statistical Tests |
|---|---|---|---|---|
| Age | Quantitative (years) | V1a (Scr) | IIT | 95% CI |
| BMI | Quantitative | V1a (Scr) | IIT | 95% CI |
| Gender | Categorical | V1a (Scr) | IIT | |
| Race | Categorical | V1a (Scr) | IIT | |
| Ethnicity | Categorical | V1a (Scr) | IIT | |
| Keloid Hx | Categorical | V1a (Scr) | IIT | |
| Smoking Hx | Categorical | V1a (Scr) | IIT | |
| Pannus Size | Categorical | V1a (Scr) | IIT | |

## **Medical History**

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Populations | Statistical Tests |
|---|---|---|---|---|
| Medical Hx | Categorical | Vla (Scr) | IIT | |

## **Concomitant Medications/Treatment**

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Populations | Statistical Tests |
|---|---|---|---|---|
| Medication | Categorical | ConMed Form | IIT | |

v.1.0; 09-Oct-2020 

## **EFFICACY ANALYSIS**

## PATIENT AND OBSERVER SCAR ASSESSMENT SCALE (POSAS; Excisions)

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Population | Statistical Tests |
|---|---|---|---|---|
| POSAS (PI) | Quantitative | V3a (D8)<br>V4a (D29)<br>V5a (D57)<br>V6a (D85) | IIT | 95% CI |
| POSAS (Subject) | Quantitative | V3a (D8)<br>V4a (D29)<br>V5a (D57)<br>V6a (D85) | IIT | 95% CI |

## TENSILE STRENGTH

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Population | Statistical Tests |
|---|---|---|---|---|
| Tensile Strength | Quantitative | V5a (D57)<br>V6a (D85) | IIT | 95% CI |

## **SAFETY ANALYSES**

## **IMMUNOGENICITY**

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Population | Statistical Tests |
|---|---|---|---|---|
| Immunogenicity | Categorical (positive / negative) | V1a (D0)<br>V3a (D8)<br>V4a (D29)<br>V5a (D57)<br>V6a (D85) | IIT | 95% CI |

## ADVERSE EVENTS

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Population | Statistical Tests |
|---|---|---|---|---|
| Adverse Events (number of subjects with and number of events): - All Adverse Events - Treatment-Emergent Adverse Events - Treatment-Related Adverse Events - Serious Adverse Events | Categorical | AE Form | SAFT | 95% CI |

v.1.0; 09-Oct-2020 

# **APPENDIX B: STATISTICAL TABLES**

| <b>14.1 SUBJECT</b> 1 | DISPOSITION | 15 |
|-----------------------|------------------------------------------------|----|
| Table 14.1.1 | Enrolment | 15 |
| Table 14.1.2 | Listing of Subject Discontinuations | 15 |
| | Subject Disposition per Visit | |
| Table 14.1.4 | Study Dates – Part A | 15 |
| 14.2 DEMOGRA | APHIC, BASELINE, AND CON-MED DETAILS | 16 |
| Table 14.2.1 | Demographics | 16 |
| Table 14.2.2 | Inclusion Criteria | 17 |
| Table 14.2.3 | Exclusion Criteria | 17 |
| Table 14.2.4 | Medical / Surgical History | 18 |
| Table 14.2.5 | Concomitant Medications/Treatment | 18 |
| 14.3 EFFICACY | Z DATA | 19 |
| | POSAS (PI Assessment, Excisions) | |
| Table 14.3.2 | POSAS (Subject Assessment, Excisions) | 20 |
| Table 14.3.4 | Tensile Strength | 21 |
| | Histology Error! Bookmark not defi | |
| 14.4 SAFETY D. | ATA | 21 |
| | Immunogenicity | |
| Table 14.4.2 | AE Profile Overview – Part A | 22 |
| Table 14.4.3 | Treatment-Emergent AEs Sorted by SOC – Part A | 22 |
| Table 14.4.4 | Treatment-Related AEs Sorted by SOC – Part A | 22 |
| Table 14.4.5 | Treatment-Emergent SAEs Sorted by SOC – Part A | 23 |
| | Treatment-Related SAEs Sorted by SOC – Part A | |

## 14.1 Subject Disposition

**Table 14.1.1 Enrolment** 

| Site | Screened | Screen Failures | Randomized | ITT | SAFT |
|-----------|----------|-----------------|------------|-----|------|
| 01 | XX | XX | xx | XX | XX |
| 02 | XX | xx | XX | XX | xx |
| 03 | XX | xx | XX | XX | xx |
| All sites | xx | xx | XX | XX | xx |

Number of Participants

**Table 14.1.2 Listing of Subject Discontinuations** 

| Subject<br>Number | Treatment<br>Group | Gender* | Age | Last<br>Visit | Primary Reason for<br>Discontinuation |
|---|---|---|---|---|---|
| #### | Active | M/F | xx | V# | xxxxxxxxxxxxxxx |
| #### | Active | M/F | XX | V# | xxxxxxxxxxxxxxxx |
| #### | Control | M/F | XX | V# | xxxxxxxxxxxxxxxx |
| #### | Active | M/F | XX | V# | xxxxxxxxxxxxxxxx |

M=Male, F=Female

Table 14.1.3 Subject Disposition per Visit

| N xx V1a (Scr) xx (xx.x%) V2a (BL/Excisions) xx (xx.x%) V3a (D8) xx (xx.x%) | Disposition of Subjects at each Study Visit | n = xx |
|---|---|---|
| V2a (BL/Excisions) xx (xx.x%) | N | xx |
| | V1a (Scr) | xx (xx.x%) |
| V3a (D8) xx (xx.x%) | V2a (BL/Excisions) | xx (xx.x%) |
| | V3a (D8) | xx (xx.x%) |
| V4a (D29) xx (xx.x%) | V4a (D29) | xx (xx.x%) |
| V5a (D57) xx (xx.x%) | V5a (D57) | xx (xx.x%) |
| V6a (D85) xx (xx.x%) | V6a (D85) | xx (xx.x%) |

Number of participants (% in parenthesis)

Table 14.1.4 Study Dates - Part A

| FPFV | LPFV | LPLV | <b>Enrollment Duration</b> | Study Duration |
|---|---|---|---|---|
| dd-mmm-yyyy | dd-mmm-yyyy | dd-mmm-yyyy | XXX | XXX |

FPFV= First Participant First Visit, LPFV= Last Participant First Visit, LPLV= Last Participant Last Visit. Enrollment duration=FPFV-LPFV+1, Study duration=FPFV-LPLV+1

v.1.0; 09-Oct-2020 

# 14.2 Demographic, Baseline, and Con-Med Details

# **Table 14.2.1 Demographics**

| | Demographics | |
|---|---|---|
| Demographics | | n = xx |
| Age | N | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) |
| | Min, Max | XX, XX |
| | Missing values | XX |
| BMI | N | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) |
| | Min, Max | XX, XX |
| | Missing values | XX |
| Gender | N | XX |
| | Male | xx (xx.x%) |
| | Female | xx (xx.x%) |
| | Missing values | XX |
| Race | N | XX |
| | American Indian or Alaska Native | xx (xx.x%) |
| | Asian | xx (xx.x%) |
| | Black or African American | xx (xx.x%) |
| | Caucasian | xx (xx.x%) |
| | Hawaiian / Pacific Islander | xx (xx.x%) |
| | Other | xx (xx.x%) |
| | Missing values | XX |
| Ethnicity | N | XX |
| | Hispanic | xx (xx.x%) |
| | Non-Hispanic | xx (xx.x%) |
| | Missing values | XX |
| Keloid/Hyp Hx | N | XX |
| | Yes | xx (xx.x%) |
| | No | xx (xx.x%) |
| | Missing values | XX |
| Smoking Hx | N | XX |
| | Non-Smoker | xx (xx.x%) |
| | Smoker | xx (xx.x%) |
| | Ex-Smoker | xx (xx.x%) |
| | Missing values | XX |
| Pannus Size | N | XX |
| | Small | xx (xx.x%) |
| | Medium | xx (xx.x%) |
| | Large | xx (xx.x%) |
| | Missing values | XX |

95% CI [xx.x, xx.x], Mean ± standard deviation. Number of Participants (% in parenthesis).

v.1.0; 09-Oct-2020 

**Table 14.2.2 Inclusion Criteria** 

| Inclusion Criteria | | n = xx |
|--------------------|-----|------------|
| Inclusion 1 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Inclusion 2 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Inclusion 3 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Inclusion 4 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Inclusion 5 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Inclusion 6 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |

Number of participants (% in parenthesis).

**Table 14.2.3 Exclusion Criteria** 

| Exclusion Criteria | | n = xx |
|--------------------|-----|------------|
| Exclusion 1 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 2 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 3 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 4 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 5 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 6 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 7 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 8 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 9 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| xclusion 10 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 11 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 12 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 13 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| xclusion 14 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 15 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 16 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |

Number of participants (% in parenthesis).

v.1.0; 09-Oct-2020 

Table 14.2.4 Medical / Surgical History

| Medical / Surgical History | n = xx |
|------------------------------------------------------|------------|
| Blood and lymphatic system disorders | xx (xx.x%) |
| 2. Cardiac/Vascular disorders | xx (xx.x%) |
| 3. Eye/Ear and labyrinth disorders | xx (xx.x%) |
| 4. Endocrine disorders | xx (xx.x%) |
| 5. Gastrointestinal/Hepatobiliary disorders | xx (xx.x%) |
| General disorders and administration site conditions | xx (xx.x%) |
| 7. Immune system disorders | xx (xx.x%) |
| 8. Infections and infestations | xx (xx.x%) |
| 9. Injury, poisoning and procedural complications | xx (xx.x%) |
| 10. Metabolism and nutrition disorders | xx (xx.x%) |
| 11. Musculoskeletal and connective tissue disorders | xx (xx.x%) |
| 12. Neoplasms benign, malignant and unspecified | xx (xx.x%) |
| 13. Nervous system disorders | xx (xx.x%) |
| 14. Psychiatric disorders | xx (xx.x%) |
| 15. Renal and urinary disorders | xx (xx.x%) |
| 16. Reproductive system and breast disorders | xx (xx.x%) |
| 17. Respiratory, thoracic and mediastinal disorders | xx (xx.x%) |
| 18. Skin and subcutaneous tissue disorders | xx (xx.x%) |
| 19. Surgical and medical procedures | xx (xx.x%) |
| 20. Allergies | xx (xx.x%) |
| 21. Other | xx (xx.x%) |

Number of Participants (% in parenthesis).

**Table 14.2.5 Concomitant Medications/Treatment** 

| Concomitant Medication/Treatment | n = xx |
|-----------------------------------------|------------|
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xx (xx.x%) |

Number of Participants (% in parenthesis).

v.1.0; 09-Oct-2020 

# 14.3 Efficacy Data

Table 14.3.1 POSAS (PI Assessment, Excisions)

| POSAS (PI | ) | | Active | Control |
|---|---|---|---|---|
| V3a (D8) | Low Tension | N | XX | XX |
| | | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | 0 | Min, Max | XX.X, XX.X | XX.X, XX.X |
| , | Opinion | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | XX.X ± XX.X [XX.X, XX.X] |
| | High Tension | | XX | XX |
| | | Mean ± SD<br>Median (P25, P75) | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Min, Max | XX.X, XX.X | xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | xx.x ± xx.x [xx.x, xx.x] |
| • | All Excisions | N | XX | XX |
| | All Excisions | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | | Min, Max | xx.x, xx.x | xx.x, xx.x |
| | Opinion | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| V4a (D29) | Low Tension | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | <b>.</b> | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | | xx.x ± xx.x [xx.x, xx.x] | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | High Tension | | XX | XX |
| | | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Median (P25, P75)<br>Min, Max | XX.X (XX.X, XX.X)<br>XX.X, XX.X | xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| | Opinion | | $XX.X \pm XX.X [XX.X, XX.X]$ | xx.x ± xx.x [xx.x, xx.x] |
| • | All Excisions | N | XX | XX |
| | All Excisions | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $XX.X \pm XX.X [XX.X, XX.X]$ |
| V5a (D57) | Low Tension | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | 0 | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | | $XX.X \pm XX.X [XX.X, XX.X]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | High Tension | | XX | XX |
| | | Mean ± SD<br>Median (P25, P75) | XX.X ± XX.X [XX.X, XX.X] | xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | XX.X ± XX.X [XX.X, XX.X] |
| • | All Excisions | N | XX | xx |
| | | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | XX.X ± XX.X [XX.X, XX.X] |
| V6a (D85) | Low Tension | N | XX | XX |
| | | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | • • • | XX.X (XX.X, XX.X) |
| | Opinion | Min, Max<br>Mean ± SD | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] | XX.X, XX.X<br>xx x + xx x [xx x xx x] |
| • | | | - | XX.X ± XX.X [XX.X, XX.X] |
| | High Tension | Mean ± SD | xx<br>xx.x ± xx.x [xx.x, xx.x] | $xx$ $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| • | All Excisions | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | | Min, Max | XX.X, XX.X | xx.x, xx.x |

N = # of excisions, 95% CI [xx.x, xx.x], Mean ± standard deviation

v.1.0; 09-Oct-2020 

Table 14.3.2 POSAS (Subject Assessment, Excisions)

| POSAS (S | ubject) | | Active | Control |
|---|---|---|---|---|
| V3a (D8) | Low Tension | N | XX | XX |
| • • | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | <b>High Tension</b> | N | XX | XX |
| | J | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | All Excisions | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | $XX.X \pm XX.X [XX.X, XX.X]$ |
| V4a (D29) | Low Tension | N | XX | XX |
| u (D20) | | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | High Tension | N | XX | XX |
| | riigii reiisioii | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | All Excisions | N | XX | XX |
| | All Excisions | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Oninion | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | XX.X ± XX.X [XX.X, XX.X] |
| VE2 (DE7) | Low Tension | N | - | |
| V3a (D31) | LOW TELISION | Mean ± SD | xx<br>xx.x ± xx.x [xx.x, xx.x] | xx<br>xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Oninion | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | XX.X ± XX.X [XX.X, XX.X] |
| | High Tension | Mean ± SD | XX | XX |
| | | Median (P25, P75) | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Min, Max | XX.X, XX.X | xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| | Oninion | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | XX.X, $XX.XXX.X \pm XX.X [XX.X, XX.X]$ |
| | | N N | | |
| | All Excisions | | XX | XX |
| | | Mean ± SD<br>Median (P25, P75) | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Min, Max | XX.X (XX.X, XX.X)<br>XX.X, XX.X | xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| | Oninion | Mean ± SD | · | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] |
| VC= (BOE) | | | XX.X ± XX.X [XX.X, XX.X] | |
| voa (D85) | Low Tension | N<br>Moon + SD | XX | XX |
| | | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Median (P25, P75) | · · · | xx.x (xx.x, xx.x) |
| | Oninion | Min, Max<br>Mean + SD | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | High Tension | | XX | XX |
| | | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | XX.X ± XX.X [XX.X, XX.X] |
| | | Median (P25, P75) | · · · | XX.X (XX.X, XX.X) |
| | <b>.</b> | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | All Excisions | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | • • | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | | Mean ± SD | | $xx.x \pm xx.x [xx.x, xx.x]$ |

N = # of excisions, 95% CI [xx.x, xx.x], Mean ± standard deviation

v.1.0; 09-Oct-2020 

**Table 14.3.4 Tensile Strength** 

| Tensile St | rength | | Active | Control |
|---|---|---|---|---|
| V5a (D57) | Low Tension | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | <b>High Tension</b> | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | All Excisions | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| V6a (D85) | Low Tension | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | <b>High Tension</b> | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | All Excisions | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |

95% CI [xx.x, xx.x] Mean ± standard deviation

# 14.4 Safety Data

**Table 14.4.1 Immunogenicity** 

| Immunoge | enicity | n = xx |
|-----------|--------------|-------------------------|
| V1a (D0) | N | XX |
| | Negative | xx (xx.x%) [xx.x, xx.x] |
| | Positive | xx (xx.x%) [xx.x, xx.x] |
| | Missing Data | XX |
| V3a (D8) | N | xx |
| | Negative | xx (xx.x%) [xx.x, xx.x] |
| | Positive | xx (xx.x%) [xx.x, xx.x] |
| | Missing Data | XX |
| V4a (D29) | N | xx |
| | Negative | xx (xx.x%) [xx.x, xx.x] |
| | Positive | xx (xx.x%) [xx.x, xx.x] |
| | Missing Data | XX |
| V5a (D57) | N | XX |
| | Negative | xx (xx.x%) [xx.x, xx.x] |
| | Positive | xx (xx.x%) [xx.x, xx.x] |
| | Missing Data | XX |
| V6a (D85) | N | XX |
| | Negative | xx (xx.x%) [xx.x, xx.x] |
| | Positive | xx (xx.x%) [xx.x, xx.x] |
| 0.50/ 015 | Missing Data | XX |

95% CI [xx.x, xx.x]

v.1.0; 09-Oct-2020 

**Table 14.4.2 AE Profile Overview – Part A** 

| | | Active (n = xx) | Control<br>(n = xx) | All (n = xx) |
|---|---|---|---|---|
| Participants with any TEAE <sup>a</sup> | Participants | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] |
| | Events | xxx | xxx | xxx |
| Participants with any TRAE <sup>b</sup> | Participants | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] |
| | Events | xxx | xxx | xxx |
| Participants with any SAE <sup>c</sup> | Participants | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] |
| | Events | xxx | xxx | xxx |
| Participants with any TRSAEd | Participants | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] |
| | Events | XXX | XXX | XXX |

95% CI [xx.x, xx.x]. aTEAE= Treatment-Emergent Adverse Events. bTRAE= Treatment-Related Adverse Events.

Table 14.4.3 Treatment-Emergent AEs Sorted by SOC – Part A

| | | Active<br>(n = xx) | | Control<br>(n = xx) | | All<br>(n = xx) | |
|---|---|---|---|---|---|---|---|
| SOC | PT | Participants | Events | Participants | Events | Participants | Events |
| Any TEAE | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| XXXXXXX | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |

95% CI [xx.x, xx.x].

Table 14.4.4 Treatment-Related AEs Sorted by SOC – Part A

| | | Active<br>(n = xx) | | Control<br>(n = xx) | | All<br>(n = xx) | |
|---|---|---|---|---|---|---|---|
| SOC | PT | Participants | Events | Participants | Events | Participants | Events |
| Any TRAE | | xx (xx.x%) [ xx.x, xx.x] | xx | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| XXXXXX | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXXX | xx (xx.x%) [ xx.x, xx.x] | xx | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |

95% CI [xx.x, xx.x].

v.1.0; 09-Oct-2020 

<sup>°</sup>SAE= Serious Adverse Events. dTRSAE= Treatment-Related Serious Adverse Events.

Table 14.4.5 Treatment-Emergent SAEs Sorted by SOC – Part A

| | | Active<br>(n = xx) | | Control<br>(n = xx) | | All<br>(n = xx) | |
|---|---|---|---|---|---|---|---|
| SOC | PT | Participants | Events | Participants | Events | Participants | Events |
| Any TESAE | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| XXXXXX | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |

95% CI [xx.x, xx.x].

Table 14.4.6 Treatment-Related SAEs Sorted by SOC – Part A

| | | Active<br>(n = xx) | | Control<br>(n = xx) | All<br>(n = xx) | | |
|---|---|---|---|---|---|---|---|
| SOC | PT | Participants | Events | Participants | Events | Participants | Events |
| Any TRSAE | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| XXXXXX | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | xx | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |

95% CI [xx.x, xx.x].

v.1.0; 09-Oct-2020 

## STATISTICAL ANALYSIS PLAN

STUDY NUMBER: SLI-C40-001
Study Part B (Abdominoplasty)

Version: v. 1.0

Date: 09-Oct-2020

Safety and Efficacy of SLI-F06 in Wound Healing and Scar Appearance in Pre-Abdominoplasty Surgical Excisions and Post-Operative Scar Appearance in Subjects Undergoing Abdominoplasty

## **Study Sponsor**

Scarless Laboratories Inc. 369 South Doheny Drive, Suite 1201 Beverly Hills, CA USA 90211

## **Clinical Research Organization**

ethica CRO Inc. 8555 Transcanada Hwy, Suite 201 Montreal, Canada H4S 1Z6 866-384-4221

#### **Confidentiality Statement**

The information contained in this document is provided in confidence. It is understood that this information will not be disclosed to others without prior agreement with the Sponsor, except to other study personnel and to the extent necessary to obtain informed consent from participating subject.

v.1.0; 09-Oct-2020 

# SAP APPROVAL SIGNATURE PAGE

The following individuals approve this version of the SLI-C40-001 Part B Statistical Analysis Plan.

| Accepted for the Sponsor – Scarless Laboratories Inc. | |
|---|---|
| Printed Name | Title |
| Signature | Date |
| Accepted for the Clinical | Research Organization - ethica CRO Inc. |
| Printed Name | Title |
| Signature | <br>Date |

v.1.0; 09-Oct-2020 

# TABLE OF CONTENTS

| SAP | APPRO | VAL SIGNATURE PAGE | 2 |
|---|---|---|---|
| TAB | LE OF C | CONTENTS | 3 |
| ABB | REVIAT | TIONS | 4 |
| 1 | INTE | RODUCTION | 5 |
| | 1.1 | Background | 5 |
| | 1.2 | Objectives | 6 |
| | 1.3 | Study Design | |
| 2 | STU | DY POPULATION | 8 |
| 3 | TRE | ATMENT ALLOCATION AND RANDOMIZATION | 8 |
| 4 | STUI | DY EVALUATIONS | 8 |
| | 4.1 | Primary Efficacy Variable | 8 |
| | 4.1.1 | | |
| | 4.2 | Secondary Efficacy Variables | |
| | 4.2.1 | POSAS (Subject Assessment) – Abdominoplasty Incisions | |
| | 4.3 | Exploratory Efficacy Variable | |
| | 4.3.1 | POSAS (PI Assessment) – Abdominoplasty Incisions, 5cm Segments | |
| | 4.3.2 | POSAS (Subject Assessment) – Abdominoplasty Incisions, 5cm Segments | |
| | 4.4 | Safety Variables | |
| | 4.4.1 | Adverse Events (AEs) | 8 |
| | 4.4.2 | Clinical Safety Laboratory Tests | 8 |
| | 4.4.3 | Immunogenicity Testing | 8 |
| | 4.4.4 | Concomitant Medications and Procedures | 8 |
| 5 | ANA | LYSIS POPULATIONS | 9 |
| | 5.1 | Populations | |
| | 5.1.1 | Intent-to-Treat (ITT) Population | |
| | 5.1.2 | Per Protocol (PP) Population | |
| | 5.1.3 | Safety (SAFT) Population | |
| 6 | SAM | PLE SIZE JUSTIFICATION | |
| 7 | | ΓISTICAL METHODS | |
| , | 7.1 | Efficacy Analyses | |
| | 7.2 | Safety Analyses | |
| | 7.3 | Adverse Events (AEs) | |
| | 7.4 | Concomitant Medications and Procedures. | |
| | 7.5 | Safety Laboratory Tests | |
| | 7.6 | Immunogenicity | |
| | 7.7 | General Statistical Considerations | |
| | 7.7.1 | Statistical Testing | |
| | 7.7.2 | Descriptive Statistics | |
| | 7.7.3 | Missing Values | |
| | 7.7.4 | Discontinuation and Drop-Outs | |
| | 7.7.5 | Multiple Comparisons | |
| | 7.7.6 | Multicenter Data | |
| | 7.7.7 | Sub-Populations Error! Bookmark not defi | |
| | 7.7.8 | Subject Disposition | |
| | 7.7.9 | Outliers | |
| | A DDEN | IDIX A: SUMMARY OF STATISTICAL TESTS | 10 |
| | | IDIX A: SUMMARY OF STATISTICAL TESTS<br>IDIX B: STATISTICAL TARI FS | 12 |

# **ABBREVIATIONS**

| AE | Adverse Event |
|---------------|-------------------------------------------------|
| BL | Baseline |
| BMI | Body Mass Index |
| CFR | U. S. Code of Federal Regulations |
| CTR | Common Treatment Response |
| CRO | Clinical Research Organization |
| DP | Drug Product |
| Excision site | A mapped area designated for a single excision. |
| eCRF | electronic Case Report Form |
| IRB | Institutional Review Board |
| ITT | Intent-to-Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PI | Principal Investigator |
| POC | Proof Of Concept |
| POSAS | Patient and Observer Scar Assessment Scale |
| PP | Per protocol |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAFT | Safety |
| SAP | Statistical Analysis Plan |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| TRAE | Treatment Related Adverse Event |
| Tx | Treatment |
| UPT | Urine Pregnancy Test |
| USP | United States Pharmacopeia |

v.1.0; 09-Oct-2020 

#### 1 INTRODUCTION

This statistical analysis plan (SAP) gives a comprehensive and detailed description of statistical techniques to be used for study SLI-C40-001. The purpose of this SAP is to ensure the credibility of the study findings by pre-specifying the statistical approaches for the analysis of study data prior to database lock. This SAP provides additional details concerning the statistical analyses outlined in the protocol. Whenever differences exist in descriptions or explanations provided in the protocol and SAP, the SAP prevails.

#### 1.1 Background

SLI-F06 is a synthetic peptide that is being developed as a treatment to promote wound healing and improve scar appearance. The amino acid sequence of SLI-F06 is derived from an endogenous human protein that has been shown in animal models to promote accelerated wound healing, reduced scarring, and increased wound tensile strength. In these same animal models, the SLI-F06 has been demonstrated to retain similar pro-migration, pro-tensile strength, and anti-fibrotic properties as the endogenous protein.

SLI-F06 drug product (DP) is a sterile lyophilized powder consisting of SLI-F06 as the active ingredient and formulation buffer components. The DP will be reconstituted in clinic with USP Water for Injection and injected intradermally along both edges of a freshly made excision to achieve a primarily local effect.

The study population will consist of healthy patients planning to undergo elective abdominoplasty. During **Part A** of this study (i.e., Phase I Safety/Proof of Concept), each subject will receive 12, 14, or 18 small or large excisions at 8 weeks or 12 weeks pre-abdominoplasty. Wounds treated with SLI-F06 or vehicle will be followed until the time of abdominoplasty when the tissue is harvested. At the completion of study Part A, subjects will enter study **Part B** where they will undergo the abdominoplasty, have the abdominoplasty incision treated with SLI-F06, and be followed for an additional 12 months.

# This SAP covers Study Part B only

v.1.0; 09-Oct-2020 

## 1.2 Objectives

The primary objectives of this study are the following:

• Assess the safety and tolerability of SLI-F06 in the treatment of abdominoplasty incisions.

Secondary objectives include, but are not limited to, the following:

- Assess the effect of SLI-F06 on post-operative abdominoplasty scar appearance.
- Assess immunogenicity effects of SLI-F06.

## 1.3 Study Design

This is a multicenter, double-blind study comparing the safety of SLI-F06 to control formulation buffer (vehicle), as well as comparing the improvement in scar appearance and wound strength. Each subject will serve as his or her own control. The study is divided into 2 parts where Part A is a Phase I safety/proof of concept study of small scars pre-abdominoplasty, and Part B is a Phase IIa study of post-abdominoplasty scars.

In **Part A** of the study (i.e., Phase I safety/proof-of-concepts. Subjects will then be randomized by side of the pannus (right or left) for treatment with SLI-F06 or formulation buffer, wound tension (high or low), and by duration of follow-up post-excisions to 12 weeks (group 1) or 8 weeks (group 2) pre-abdominoplasty. Excision mapping and number of excisions will be determined by size of pannus as follows:

- Small pannus: 6 low tension and 6 high tension wounds will (12 wounds/subject).
- Medium pannus: 6 low tension and 8 high tension wounds will (14 wounds/subject).
- Large pannus: 8 low tension and 10 high tension wounds (18 wounds/subject).

Following completion of the follow-up period, the entire abdominoplasty site will be harvested and sent for analyses of histopathology and tensile strength.

In **Part B** of the study (i.e., Phase IIa), <u>ALL</u> subjects who complete Part A will be randomly assigned to receive injections of SLI-F06 along one half (left or right) of the abdominoplasty incision and control injections along the other half. The subject will undergo routine wound care and will attend study follow-up visits following abdominoplasty at Day 8 and at Months 1, 2, 3, 6, 9, and 12.

v.1.0; 09-Oct-2020 

## **STUDY SUMMARY**

| | | Part A (P | hase I Safety/P | roof of C | Concept) | | | | | Part l | B (Phase | IIa) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | 1a | 2a | 3a | 4a | 5a | 6a | 1b | 2b | SR | 3b | 4b | 5b | 6b | 7b | 8b |
| Assessment and Procedures | Screening<br>Period | Excisions | Suture<br>Removal | | | | Abdomin-<br>oplasty | | Suture<br>Removal | | | | | | |
| Assessment and Frocedures | D -30<br>to 0 | D1 | D8<br>± 1d | D29<br>± 2d | D57<br>± 3d | D85<br>± 3d | D0 | D8<br>± 1d | PI<br>Discretion | M1<br>± 3d | M2<br>± 7d | M3<br>± 14d | M6<br>± 14d | M9<br>± 14d | M12<br>± 14d |
| Informed Consent | X | | | | | | | | | | | | | | |
| Inc/Excl Criteria | X | | | | | | | | | | | | | | |
| Medical/Surgical History | X | | | | | | | | | | | | | | |
| Physical Exam | X | | | | | | | | | | | | | | |
| Urine Pregnancy Test <sup>1</sup> | X | X 1 | | | | | X | | | | | X | X | X | X |
| Abdominoplasty Area Assessment & selection of Pannus Map size | X | | | | | | | | | | | | | | |
| Immunogenicity sampling | X | | X | X | X | X | | X | | X | X | X | X | X | X |
| Safety Laboratory Testing <sup>2</sup> | X 2 | | | X | Group 2 | Group 1 | | | | X | | | | | X |
| Photography <sup>3</sup> | | X 3 | X 3 | X | X | X | | | | X | X | X | X | X | X |
| Randomization | | X | | | | | X | | | | | | | | |
| Excisions | | X | | | | | | | | | | | | | |
| IP Injections | | X | | | | | X | | | | | | | | |
| Abdominoplasty/ Tissue<br>Harvesting | | | | | | | X | | | | | | | | 1 |
| Suture removal | | | X | | | | | | X | | | | | | |
| POSAS grading | | | Post-removal of sutures | X | X | X | | | | X | X | X | X | X | X |
| AE Assessment | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Group 1; 12 week assessment | | | | | | | | | | | - | | | | |
| Exit from Part A / Start of Part B | | | | | | X | | | | | | | | | |
| Group 2; 8 week assessment <sup>4</sup> | | | | | | | | | | | | | | | |
| Exit from Part A / Start of Part B | | | | | X | | | | | | | | | | |

<sup>1</sup> UPT if female of childbearing potential and if last UPT performed >7 days of V2a.

v.1.0; 09-Oct-2020 

<sup>2</sup> Safety laboratory results to be reviewed by the PI prior to excisions in order to confirm absence of any health condition(s) that would make the subject inappropriate for study entry.

<sup>3</sup> Day 1 photography occurs prior to excisions and following closure of all excisions, and Day 8 photography occurs pre- and post-removal of sutures.

 $<sup>\</sup>textbf{4} \ \text{Only } \textbf{currently enrolled} \ \text{participants who cannot be moved from group 2 to group 1 will remain in group 2}$ 

#### 2 STUDY POPULATION

Healthy adult subjects presenting for abdominoplasty surgery will be enrolled and randomized. The full description of the inclusion and exclusion criteria is found in Section 5 of the study protocol.

#### 3 TREATMENT ALLOCATION AND RANDOMIZATION

One side of the abdominoplasty incision will be treated with SLI-F06 (i.e., left side or right side) and the other side of the incision will be treated with vehicle.

#### 4 STUDY EVALUATIONS

## 4.1 Primary Efficacy Variable

## 4.1.1 POSAS (PI Assessment) – Abdominoplasty Incisions

The Patient and Observer Scar Assessment Scale (POSAS) will be used to assess the various parameters of the abdominoplasty incision. At each observation time point, the <u>PI</u> will grade each scar using the "Observer Scale" of the POSAS.

## 4.2 Secondary Efficacy Variables

## 4.2.1 POSAS (Subject Assessment) – Abdominoplasty Incisions

Subjects will grade the abdominoplasty scar using the "Patient Scale" criteria of the POSAS.

#### 4.3 Exploratory Efficacy Variable

## 4.3.1 POSAS (PI Assessment) – Abdominoplasty Incisions, 5cm Segments

The Patient and Observer Scar Assessment Scale (POSAS) will be used to assess the various parameters of the abdominoplasty incision at 5cm intervals. At each observation time point, the <u>PI</u> will grade each scar using the "Observer Scale" of the POSAS.

## 4.3.2 POSAS (Subject Assessment) – Abdominoplasty Incisions, 5cm Segments

The Patient and Observer Scar Assessment Scale (POSAS) will be used to assess the various parameters of the abdominoplasty incision at 5cm intervals. At each observation time point, the subject will grade each scar using the "Observer Scale" of the POSAS.

#### 4.4 Safety Variables

#### 4.4.1 Adverse Events (AEs)

The Treating Investigator will assess AEs and record details of seriousness, severity, duration, and action taken with the study device, and relationship to the study device.

#### 4.4.2 Clinical Safety Laboratory Tests

Standard clinical laboratory analyses (CBC/Diff, chemistry) will be conducted on blood samples collected at V3b (M1) and V8b (M12). Clinically significant results, in the opinion of the PI, will be reported as AEs.

## 4.4.3 Immunogenicity Testing

Immunogenicity analyses will be conducted at V2b (Day 8), V3b (M1), V4b (M2), V5b (M3), V6b (M6), V7b (M9), and V8b (M12).

#### 4.4.4 Concomitant Medications and Procedures

Any medication or procedure (including OTC preparations) that the subject takes during the study protocol period will be considered concomitant medication and will recorded.

v.1.0; 09-Oct-2020 

#### 5 ANALYSIS POPULATIONS

## 5.1 Populations

## 5.1.1 Intent-to-Treat (ITT) Population

The ITT population will be the primary population for efficacy and safety analyses and will consist of all randomized subjects who received at least one injection of IP and provided at least one post-baseline evaluation, and will be analyzed in the treatment group they were allocated.

#### 5.1.2 Per Protocol (PP) Population

A per-protocol (PP) population will neither be identified nor analyzed.

## 5.1.3 Safety (SAFT) Population

The SAFT population will be used for safety analysis and will consist of all randomized subjects who received one injection of IP, and will be analyzed as per the treatment actually received.

#### 6 SAMPLE SIZE JUSTIFICATION

This is a Phase IIa study and a formal sample size justification is not required. It is the opinion of the Sponsor that a total of 25 subjects will be sufficient to achieve the objectives of the study.

#### 7 STATISTICAL METHODS

## 7.1 Efficacy Analyses

Efficacy analyses will be conducted on an intent-to-treat (ITT) basis.

For categorical parameters, the number and percentage of subjects/observations in each category will be presented. The denominator will be based on the number of subjects/observations appropriate for the purpose of analysis. For continuous parameters, descriptive statistics will include n (number of subjects or observations), mean, standard deviation, median, and range.

Comparisons between treatment groups will be based on 95% confidence intervals.

## 7.2 Safety Analyses

Safety analysis will be conducted on the Safety Population (SAFT), by tabulations of AEs, safety laboratory parameters and immunogenicity outcomes.

Subjects will be followed for AEs (local and systemic) throughout the study. Events specific to treatment sites will be recorded per side to allow comparison of study treatments.

#### 7.3 Adverse Events (AEs)

Safety outcomes will be incidence rate of AEs, including SAEs, types of AEs and relationship to study treatment (i.e., Treatment-Emergent Adverse Events [TEAEs]; Treatment-Related-Adverse Events [TRAEs]). TEAEs will include all reported AE since the time of informed consent. TRAEs will include all reported AEs that were deemed by the Investigator to be related or not-related to study treatment.

Safety data will be tabulated with descriptive group statistics (mean, standard deviation, minimum, maximum). Severity and relationship to study treatment will be assessed.

AEs will be coded using MedDRA. These events, irrespective of relationship to study medication, will be summarized by treatment groups, MedDRA system organ class (SOC) and MedDRA preferred term (PT). The number of subjects reporting an AE, the number of AEs, and percentages of subjects in each category will be summarized. AEs by severity and relationship to study will be summarized in a similar way. Serious AEs will be summarized separately. Specifically, the

v.1.0; 09-Oct-2020 

following AE incidence tables will be provided:

- Treatment-Emergent AEs: Sorted By SOC and PT
- Treatment-Related AEs: Sorted By SOC and PT
- Treatment-Emergent SAEs: Sorted By SOC and PT
- Treatment-Related SAEs: Sorted By SOC and PT

AE incidence rates with exact 95% confidence intervals will be calculated for each safety variable; confidence intervals will be used to confirm whether distribution of subjects with events is homogeneous between the treatment groups.

#### 7.4 Concomitant Medications and Procedures

Descriptive statistics (i.e., frequency and percent) will be calculated for each treatment group.

#### 7.5 Safety Laboratory Tests

Determination of clinical significance for all out-of-range laboratory values will be made by each PI, and Adverse Event reports will be generated as necessary.

## 7.6 Immunogenicity

Changes from baseline in immunogenicity outcomes will be summarized with descriptive statistics and text, as appropriate.

#### 7.7 General Statistical Considerations

## 7.7.1 Statistical Testing

For specific information regarding the statistical tests to be used in this study, please refer to Appendix A: Summary of Statistical Tests. Comparisons between treatment groups will be based on 95% confidence intervals.

#### 7.7.2 Descriptive Statistics

Descriptive statistics (i.e., frequency and percent) will be calculated for each treatment group. Quantitative variables will be presented by way of number of observations, number of missing values, mean, standard deviation, extreme values (minimum and maximum), median, and 95% confidence internals. Categorical data will be presented by way of number of observations, number of missing values, and for each observed category, the number of occurrences and its corresponding percentage, and 95% confidence internals.

#### 7.7.3 Missing Values

Missing data will not be imputed. Data will be analyzed as observed.

#### 7.7.4 Discontinuation and Drop-Outs

Dropouts will not be replaced. All available data from dropouts will be included in the ITT analysis.

#### 7.7.5 Multiple Comparisons

No methods will be used to accommodate multiplicity (unless otherwise specified).

#### 7.7.6 Multicenter Data

The data will be pooled across centers for analysis. Additionally, data for each center will be provided in data listings.

v.1.0; 09-Oct-2020 

## 7.7.7 Subject Disposition

A tabulation of subject disposition will be provided which will include the numbers of subjects who enter, complete, and discontinue the study. The reasons for discontinuation will be included.

## 7.7.8 Outliers

No method to process outliers will be used. Data will be analyzed as reported in the database.

v.1.0; 09-Oct-2020 

# APPENDIX A: SUMMARY OF STATISTICAL TESTS

## STUDY DISPOSITION

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Populations | Statistica<br>1 Tests |
|---|---|---|---|---|
| Subject discontinuations | Listing: - Last Visit - Reason for discontinuing | Exit Form | IIT | |
| Primary Reason for discontinuations | Categorical | Exit Form | IIT | |
| Disposition at each Visit | Frequency of subjects attending visit | All Visits | IIT | |
| Study dates | <ul> <li>FPFV</li> <li>LPFV</li> <li>LPLV</li> <li>Enrolment duration</li> <li>Study duration</li> </ul> | All Visits | IIT | |

## **BASELINE CHARACTERISTICS**

## **Demographics**

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Populations | Statistical Tests |
|---|---|---|---|---|
| Age | Quantitative (years) | V1a (Scr) | IIT | 95% CI |
| BMI | Quantitative | V1a (Scr) | IIT | 95% CI |
| Gender | Categorical | V1a (Scr) | IIT | |
| Race | Categorical | V1a (Scr) | IIT | |
| Ethnicity | Categorical | V1a (Scr) | IIT | |
| Keloid Hx | Categorical | V1a (Scr) | IIT | |
| Smoking Hx | Categorical | V1a (Scr) | IIT | |
| Pannus Size | Categorical | V1a (Scr) | IIT | |

## **Medical History**

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Populations | Statistical Tests |
|---|---|---|---|---|
| Medical Hx | Categorical | Vla (Scr) | IIT | |

## **Concomitant Medications/Treatment**

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Populations | Statistical Tests |
|---|---|---|---|---|
| Medication | Categorical | ConMed Form | IIT | |

v.1.0; 09-Oct-2020 

## **EFFICACY ANALYSIS**

## PATIENT AND OBSERVER SCAR ASSESSMENT SCALE (POSAS; Excisions)

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Population | Statistical Tests |
|---|---|---|---|---|
| POSAS (PI) | Quantitative | V3b (M1)<br>V4b (M2)<br>V5b (M3)<br>V6b (M6)<br>V7b (M9)<br>V8b (M12) | IIT | 95% CI |
| POSAS (Subject) | Quantitative | V3b (M1)<br>V4b (M2)<br>V5b (M3)<br>V6b (M6)<br>V7b (M9)<br>V8b (M12) | IIT | 95% CI |
| POSAS (PI; 5cm<br>Segment) | Quantitative | V5b (M3)<br>V6b (M6)<br>V7b (M9)<br>V8b (M12) | IIT | 95% CI |
| POSAS (Subject;<br>5cm Segment) | Quantitative | V5b (M3)<br>V6b (M6)<br>V7b (M9)<br>V8b (M12) | IIT | 95% CI |

## **SAFETY ANALYSES**

## **IMMUNOGENICITY**

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Population | Statistical Tests |
|---|---|---|---|---|
| Immunogenicity | Categorical (positive / negative) | V2b (D8)<br>V3b (M1)<br>V4b (M2)<br>V5b (M3)<br>V6b (M6)<br>V7b (M9)<br>V8b (M12) | IIT | 95% CI |

## ADVERSE EVENTS

| Variable | Туре | Visits /<br>CRF Section | Analyzed<br>Population | Statistical Tests |
|---|---|---|---|---|
| Adverse Events (number of subjects with and number of events): - All Adverse Events - Treatment-Emergent Adverse Events - Treatment-Related Adverse Events - Serious Adverse Events | Categorical | AE Form | SAFT | 95% CI |

v.1.0; 09-Oct-2020 
## **APPENDIX B: STATISTICAL TABLES**

| 14.1 SUBJECT | DISPOSITION | 15 |
|---|---|---|
| Table 14.1.1 | Enrolment | 15 |
| Table 14.1.2 | Listing of Subject Discontinuations | 15 |
| Table 14.1.3 | Subject Disposition per Visit | 15 |
| Table 14.1.4 | Study Dates – Part B | 15 |
| 14.2 DEMOGR | APHIC, BASELINE, AND CON-MED DETAILS | 16 |
| | Demographics | |
| Table 14.2.2 | Inclusion Criteria | 17 |
| Table 14.2.3 | Exclusion Criteria | 17 |
| Table 14.2.4 | Medical / Surgical History | 18 |
| Table 14.2.5 | Concomitant Medications/Treatment | 18 |
| 14.3 EFFICACY | Y DATA | 19 |
| Table 14.3.1 | POSAS (PI Assessment, Abdominoplasty, Full Scar) | 19 |
| Table 14.3.2 | POSAS (Subject Assessment, Abdominoplasty, Full Scar) | 20 |
| Table 14.3.3 | POSAS (PI Assessment, Abdominoplasty, 5cm Segments) | 21 |
| Table 14.3.4 | POSAS (Subject Assessment, Abdominoplasty, 5cm Segments) | 23 |
| 14.4 SAFETY D | ATA | 25 |
| | Immunogenicity | |
| | AE Profile Overview – Part B. | |
| Table 14.4.3 | Treatment-Emergent AEs Sorted by SOC – Part B | 26 |
| | Treatment-Related AEs Sorted by SOC – Part B | |
| Table 14.4.5 | Treatment-Emergent SAEs Sorted by SOC – Part B | 27 |
| | Treatment-Related SAEs Sorted by SOC – Part B | |

#### 14.1 Subject Disposition

**Table 14.1.1 Enrolment** 

| Site | Screened | Screen Failures | Randomized | PP | ITT | SAFT |
|-----------|----------|-----------------|------------|----|-----|------|
| 01 | XX | XX | xx | XX | XX | XX |
| 02 | XX | xx | XX | XX | XX | xx |
| 03 | XX | xx | XX | XX | XX | xx |
| All sites | xx | xx | XX | XX | XX | xx |

Number of Participants

**Table 14.1.2 Listing of Subject Discontinuations** 

| Subject | Treatment | Gender* | Age | Last | Primary Reason for |
|---------|-----------|---------|-----|-------|--------------------|
| Number | Group | | | Visit | Discontinuation |
| #### | Active | M/F | XX | V# | xxxxxxxxxxxxxxxx |
| #### | Active | M/F | XX | V# | xxxxxxxxxxxxxxxx |
| #### | Control | M/F | XX | V# | xxxxxxxxxxxxxxxx |
| #### | Active | M/F | XX | V# | XXXXXXXXXXXXXXXXXX |

M=Male, F=Female

Table 14.1.3 Subject Disposition per Visit

| Disposition of Subjects at each Study Visit | n = xx |
|---------------------------------------------|------------|
| N | XX |
| V1b (Abdominoplasty) | xx (xx.x%) |
| V2b (D8) | xx (xx.x%) |
| V3b (M1) | xx (xx.x%) |
| V4b (M2) | xx (xx.x%) |
| V5b (M3) | xx (xx.x%) |
| V6b (M6) | xx (xx.x%) |
| V7b (M9) | xx (xx.x%) |
| V8b (M12) | xx (xx.x%) |

Number of Participants (% in parenthesis)

**Table 14.1.4 Study Dates – Part B** 

| FPFV | LPFV | LPLV | <b>Enrollment Duration</b> | Study Duration |
|---|---|---|---|---|
| dd-mmm-yyyy | dd-mmm-yyyy | dd-mmm-yyyy | XXX | XXX |

FPFV= First Participant First Visit, LPFV= Last Participant First Visit, LPLV= Last Participant Last Visit. Enrollment duration=FPFV-LPFV+1, Study duration=FPFV-LPLV+1

v.1.0; 09-Oct-2020 

#### 14.2 Demographic, Baseline, and Con-Med Details

### **Table 14.2.1 Demographics**

| | Demographies | |
|---|---|---|
| Demographics | | n = xx |
| Age | N | xx |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) |
| | Min, Max | XX, XX |
| | Missing values | XX |
| BMI | N | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) |
| | Min, Max | XX, XX |
| | Missing values | XX |
| Gender | N | XX |
| | Male | xx (xx.x%) |
| | Female | xx (xx.x%) |
| | Missing values | XX |
| Race | N | XX |
| | American Indian or Alaska Native | xx (xx.x%) |
| | Asian | xx (xx.x%) |
| | Black or African American | xx (xx.x%) |
| | Caucasian | xx (xx.x%) |
| | Hawaiian / Pacific Islander | xx (xx.x%) |
| | Other | xx (xx.x%) |
| | Missing values | XX |
| Ethnicity | N | XX |
| | Hispanic | xx (xx.x%) |
| | Non-Hispanic | xx (xx.x%) |
| | Missing values | XX |
| Keloid/Hyp Hx | N | XX |
| | Yes | xx (xx.x%) |
| | No | xx (xx.x%) |
| | Missing values | XX |
| Smoking Hx | N | XX |
| | Non-Smoker | xx (xx.x%) |
| | Smoker | xx (xx.x%) |
| | Ex-Smoker | xx (xx.x%) |
| | Missing values | xx |
| Pannus Size | N | XX |
| | Small | xx (xx.x%) |
| | Medium | xx (xx.x%) |
| | Large | xx (xx.x%) |
| | Missing values | xx |

95% CI [xx.x, xx.x], Mean ± standard deviation. Number of Participants (% in parenthesis).

v.1.0; 09-Oct-2020 

**Table 14.2.2 Inclusion Criteria** 

| Inclusion Criteria | | n = xx |
|--------------------|-----|------------|
| Inclusion 1 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Inclusion 2 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Inclusion 3 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Inclusion 4 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Inclusion 5 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Inclusion 6 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |

Number of Participants (% in parenthesis).

**Table 14.2.3 Exclusion Criteria** 

| <b>Exclusion Criteria</b> | | n = xx |
|---------------------------|-----|------------|
| Exclusion 1 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 2 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 3 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 4 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 5 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 6 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 7 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 8 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 9 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 10 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 11 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 12 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 13 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 14 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 15 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |
| Exclusion 16 | No | xx (xx.x%) |
| | Yes | xx (xx.x%) |

Number of Participants (% in parenthesis).

v.1.0; 09-Oct-2020 

Table 14.2.4 Medical / Surgical History

| Medical / Surgical History | n = xx |
|---------------------------------------------------------|------------|
| Blood and lymphatic system disorders | xx (xx.x%) |
| 2. Cardiac/Vascular disorders | xx (xx.x%) |
| 3. Eye/Ear and labyrinth disorders | xx (xx.x%) |
| 4. Endocrine disorders | xx (xx.x%) |
| 5. Gastrointestinal/Hepatobiliary disorders | xx (xx.x%) |
| 6. General disorders and administration site conditions | xx (xx.x%) |
| 7. Immune system disorders | xx (xx.x%) |
| 8. Infections and infestations | xx (xx.x%) |
| 9. Injury, poisoning and procedural complications | xx (xx.x%) |
| 10. Metabolism and nutrition disorders | xx (xx.x%) |
| 11. Musculoskeletal and connective tissue disorders | xx (xx.x%) |
| 12. Neoplasms benign, malignant and unspecified | xx (xx.x%) |
| 13. Nervous system disorders | xx (xx.x%) |
| 14. Psychiatric disorders | xx (xx.x%) |
| 15. Renal and urinary disorders | xx (xx.x%) |
| 16. Reproductive system and breast disorders | xx (xx.x%) |
| 17. Respiratory, thoracic and mediastinal disorders | xx (xx.x%) |
| 18. Skin and subcutaneous tissue disorders | xx (xx.x%) |
| 19. Surgical and medical procedures | xx (xx.x%) |
| 20. Allergies | xx (xx.x%) |
| 21. Other | xx (xx.x%) |

Number of Participants (% in parenthesis).

**Table 14.2.5 Concomitant Medications/Treatment** 

| Concomitant Medication/Treatment | n = xx |
|-----------------------------------------|------------|
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xx (xx.x%) |

Number of Participants (% in parenthesis).

v.1.0; 09-Oct-2020 

### 14.3 Efficacy Data

Table 14.3.1 POSAS (PI Assessment, Abdominoplasty, Full Scar)

| , | | | |
|---|---|---|---|
| POSAS (PI | ) | Active | Control |
| V3b (M1) | N | XX | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| V4b (M2) | N | XX | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| V5b (M3) | N | XX | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| V6b (M6) | N | XX | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| V7b (M9) | N | XX | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| V8b (M12) | N | XX | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |

95% CI [xx.x, xx.x] Mean ± standard deviation

v.1.0; 09-Oct-2020 

Table 14.3.2 POSAS (Subject Assessment, Abdominoplasty, Full Scar)

| POSAS (Si | ubject) | Active | Control |
|---|---|---|---|
| V3b (M1) | N | XX | XX |
| () | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | Min, Max | | xx.x, xx.x |
| | | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| V4b (M2) | N | xx | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | | XX.X, XX.X |
| | Opinion | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| V5b (M3) | N | xx | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| V6b (M6) | N | xx | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | | XX.X, XX.X | XX.X, XX.X |
| | Opinion | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| V7b (M9) | N | xx | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| V8b (M12) | N | xx | XX |
| | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x(xx.x, xx.x) |
| | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |

v.1.0; 09-Oct-2020 

Table 14.3.3 POSAS (PI Assessment, Abdominoplasty, 5cm Segments)

| POSAS (F | 기) | | Active | Control |
|---|---|---|---|---|
| V5b (M3) | Seg 1 | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | Oninion | Min, Max<br>Mean ± SD | XX.X, XX.X | XX.X, XX.X |
| | Seg 2 | N | xx.x ± xx.x [xx.x, xx.x]<br>xx | xx.x ± xx.x [xx.x, xx.x]<br>xx |
| | | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | Seg 3 | N<br>Mean ± SD | XX × | XX |
| | | Median (P25, P75) | XX.X ± XX.X [XX.X, XX.X]<br>xx x (xx x xx x) | xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | Seg 4 | N | XX | XX |
| | | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | Opinion | Min, Max<br>Mean ± SD | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] |
| | Seg 5 | N | XX | XX |
| | - <b>J</b> - | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | , , , | xx.x (xx.x, xx.x) |
| | <b>2</b> · · | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | Seg 6 | N<br>Mean ± SD | xx<br>xx.x ± xx.x [xx.x, xx.x] | xx<br>xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | Q1/2/3/4/5/6 | | $xx.x \pm xx.x [xx.x, xx.x]$ | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | Oninion | Min, Max<br>Mean + SD | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] | XX.X, XX.X |
| /6b (M6) | | Mean ± SD<br>N | XX.X ± XX.X [XX.X, XX.X] XX | xx.x ± xx.x [xx.x, xx.x]<br>xx |
| (IIIO) | g . | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | | XX.X ± XX.X [XX.X, XX.X] | xx.x ± xx.x [xx.x, xx.x] |
| | Seg 2 | N<br>Mean ± SD | XX | XX<br>vv v + vv v [vv v vv v] |
| | | Median (P25, P75) | xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x) | xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | | XX.X ± XX.X [XX.X, XX.X] | xx.x ± xx.x [xx.x, xx.x] |
| | Seg 3 | N | XX | XX |
| | | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75)<br>Min, Max | xx.x (xx.x, xx.x)<br>xx.x, xx.x | XX.X (XX.X, XX.X) |
| | Opinion | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] |
| | Seg 4 | N | XX | XX |
| | • | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | O: : | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion<br>Sea 5 | Mean ± SD<br>N | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | Seg 5 | N<br>Mean ± SD | xx<br>xx.x ± xx.x [xx.x, xx.x] | $xx$ $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Seg 6 | N | XX | XX |
| | | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | Opinion | Min, Max<br>Mean ± SD | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] |
| | Q1/2/3/4/5/6 | | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Median (P25, P75) | XX.X (XX.X, XX.X) | XX.X (XX.X, XX.X) |
| | | Min, Max | xx.x, xx.x | xx.x, xx.x |
| | Opinion | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |

v.1.0; 09-Oct-2020 

Table 14.3.3 POSAS (PI Assessment, Abdominoplasty, 5cm Segments) con't

| POSAS (PI | ) | | Active | Control |
|---|---|---|---|---|
| V7b (M9) | Seg 1 | N | XX | XX |
| | | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | Oninion | Min, Max<br>Mean ± SD | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] |
| | Seg 2 | N N | XX | XX |
| | <b>J</b> | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | • • • | xx.x (xx.x, xx.x) |
| | 0 | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | Seg 3 | N<br>Mean ± SD | $XX$ $XX.X \pm XX.X [XX.X, XX.X]$ | $XX$ $XX.X \pm XX.X [XX.X, XX.X]$ |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | | Min, Max | xx.x, xx.x | XX.X, XX.X |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | Seg 4 | N | XX | XX |
| | | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Median (P25, P75)<br>Min, Max | XX.X (XX.X, XX.X)<br>XX.X, XX.X | XX.X (XX.X, XX.X) |
| | Opinion | | xx.x ± xx.x [xx.x, xx.x] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] |
| | Seg 5 | N | XX | XX |
| | _ | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | Oninian | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion Seg 6 | Mean ± SD<br>N | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x]<br>xx |
| | Jeg v | Mean ± SD | xx<br>xx.x ± xx.x [xx.x, xx.x] | xx<br>xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | Q1/2/3/4/5/6 | | xx.x ± xx.x [xx.x, xx.x] | XX.X ± XX.X [XX.X, XX.X] |
| | | Median (P25, P75)<br>Min, Max | xx.x (xx.x, xx.x)<br>xx.x, xx.x | XX.X (XX.X, XX.X)<br>XX.X, XX.X |
| | Opinion | | xx.x ± xx.x [xx.x, xx.x] | $XX.X \pm XX.X [XX.X, XX.X]$ |
| /8b (M12) | | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | Oninian | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion Seg 2 | Mean ± SD<br>N | xx.x ± xx.x [xx.x, xx.x] | XX.X ± XX.X [XX.X, XX.X] XX |
| | Oeg 2 | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | | xx.x ± xx.x [xx.x, xx.x] | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | Seg 3 | N<br>Mean ± SD | XX | XX |
| | | Median (P25, P75) | xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x) | xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Seg 4 | N<br>M | XX | XX |
| | | | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Mean ± SD | | |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Opinion | Median (P25, P75)<br>Min, Max | | |
| | Opinion Seg 5 | Median (P25, P75)<br>Min, Max | xx.x (xx.x, xx.x)<br>xx.x, xx.x | xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| | | Median (P25, P75) Min, Max Mean ± SD N Mean ± SD | XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X] | xx.x (xx.x, xx.x)<br>xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) Min, Max Mean ± SD N Mean ± SD Median (P25, P75) | XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X) | xx.x (xx.x, xx.x)<br>xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x]<br>xx.x ± xx.x [xx.x, xx.x] |
| | Seg 5 | Median (P25, P75) Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max | XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X)<br>XX.X, XX.X | xx.x (xx.x, xx.x)<br>xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x)<br>xx.x (xx.x, xx.x) |
| | Seg 5 Opinion | Median (P25, P75) Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD | XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X] | XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X] |
| | Seg 5 | Median (P25, P75) Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max | XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X ± XX.X [XX.X, XX.X] | xx.x (xx.x, xx.x)<br>xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x)<br>xx.x (xx.x, xx.x)<br>xx.x ± xx.x [xx.x, xx.x]<br>xx.x ± xx.x [xx.x, xx.x] |
| | Seg 5 Opinion | Median (P25, P75) Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N | XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X] | XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X] |
| | Seg 5 Opinion | Median (P25, P75) Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD | XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X] | xx.x (xx.x, xx.x)<br>xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x)<br>xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x] |
| | Opinion Seg 6 Opinion | Median (P25, P75) Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD | XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] | xx.x (xx.x, xx.x)<br>xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x)<br>xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x)<br>xx.x (xx.x, xx.x)<br>xx.x (xx.x, xx.x) |
| | Opinion Seg 6 | Median (P25, P75) Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD Median (P25, P75) Min, Max Mean ± SD Mean ± SD | XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] | XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 6 Opinion | Median (P25, P75) Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD | XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] | XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] |

v.1.0; 09-Oct-2020 

Table 14.3.4 POSAS (Subject Assessment, Abdominoplasty, 5cm Segments)

| POSAS (S | | | Active | Control |
|---|---|---|---|---|
| <sup>7</sup> 5b (M3) | Seg 1 | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | , , | XX.X (XX.X, XX.X) |
| | Ominian | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Seg 2 | Mean ± SD<br>N | XX.X ± XX.X [XX.X, XX.X] | xx.x ± xx.x [xx.x, xx.x]<br>xx |
| | Seg 2 | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | Seg 3 | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | Opinion | Min, Max<br>Mean ± SD | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] | xx.x, xx.x<br>$xx.x \pm xx.x [xx.x, xx.x]$ |
| | Seg 4 | N N | XX | XX |
| | oog . | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Seg 5 | N | XX | XX |
| | | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Median (P25, P75)<br>Min, Max | XX.X (XX.X, XX.X)<br>XX.X, XX.X | XX.X (XX.X, XX.X) |
| | Opinion | | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] |
| | Seg 6 | N N | XX | XX |
| | g - | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | Q1/2/3/4/5/6 | | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | Opinion | Min, Max<br>Mean ± SD | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] | xx.x, xx.x<br>$xx.x \pm xx.x [xx.x, xx.x]$ |
| /6b (M6) | | N | XX | XX |
| 7 O.D. (1810) | ocg i | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | xx.x, xx.x |
| | Opinion | | $XX.X \pm XX.X [XX.X, XX.X]$ | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | Seg 2 | N | XX | XX |
| | | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | Oninion | Min, Max<br>Mean ± SD | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] |
| | Seg 3 | N | XX | XX |
| | 9 - | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | Seg 4 | N<br>Marara 4 OD | XX | XX |
| | | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Median (P25, P75)<br>Min, Max | | XX.X (XX.X, XX.X) |
| | Opinion | Mean ± SD | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] | xx.x, xx.x<br>$xx.x \pm xx.x [xx.x, xx.x]$ |
| | Seg 5 | N | XX | XX |
| | - <b>J</b> - | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | $XX.X \pm XX.X [XX.X, XX.X]$ |
| | Seg 6 | N<br>Marara 4 OD | XX | XX |
| | | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | Oninion | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion Q1/2/3/4/5/6 | Mean ± SD<br>Mean ± SD | xx.x ± xx.x [xx.x, xx.x]<br>xx.x ± xx.x [xx.x, xx.x] | $\begin{array}{c} xx.x \pm xx.x [xx.x, xx.x] \\ xx.x \pm xx.x [xx.x, xx.x] \end{array}$ |
| | Q 11213141310 | Median (P25, P75) | | XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | | | xx.x ± xx.x [xx.x, xx.x] | |

v.1.0; 09-Oct-2020 

Table 14.3.3 POSAS (PI Assessment, Abdominoplasty, 5cm Segments) con't

| POSAS (Si | ubject) | | Active | Control |
|---|---|---|---|---|
| V7b (M9) | Seg 1 | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | The state of the s | xx.x (xx.x, xx.x) |
| | 0 | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | Seg 2 | N<br>Maari I CD | XX | XX |
| | | Mean ± SD<br>Median (P25, P75) | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | | Min, Max | XX.X (XX.X, XX.X)<br>XX.X, XX.X | XX.X (XX.X, XX.X)<br>XX.X, XX.X |
| | Opinion | | xx.x ± xx.x [xx.x, xx.x] | XX.X ± XX.X [XX.X, XX.X] |
| | Seg 3 | N | XX | XX |
| | 0090 | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | XX.X ± XX.X [XX.X, XX.X] |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Seg 4 | N | XX | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | | xx.x (xx.x, xx.x) |
| | Oninia- | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | Seg 5 | N<br>Mean ± SD | xx<br>xx.x ± xx.x [xx.x, xx.x] | xx<br>xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | Opinion | Mean ± SD | XX.X ± XX.X [XX.X, XX.X] | XX.X ± XX.X [XX.X, XX.X] |
| | Seg 6 | N | XX | XX |
| | _ | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Q1/2/3/4/5/6 | | xx.x ± xx.x [xx.x, xx.x] | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | The state of the s | XX.X (XX.X, XX.X) |
| | Oninian | Min, Max | XX.X, XX.X | XX.X, XX.X |
| V8b (M12) | Opinion<br>Soc 1 | Mean ± SD<br>N | xx.x ± xx.x [xx.x, xx.x] | XX.X ± XX.X [XX.X, XX.X] XX |
| VOD (W112) | Seg i | Mean ± SD | xx.x ± xx.x [xx.x, xx.x] | xx.x ± xx.x [xx.x, xx.x] |
| | | Median (P25, P75) | | XX.X (XX.X, XX.X) |
| | | Min, Max | xx.x, xx.x | xx.x, xx.x |
| | Opinion | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | Seg 2 | N | xx | XX |
| | | Mean ± SD | $xx.x \pm xx.x [xx.x, xx.x]$ | $xx.x \pm xx.x [xx.x, xx.x]$ |
| | | Median (P25, P75) | xx.x (xx.x, xx.x) | |
| | | | 10/1/ 10/1/ | xx.x (xx.x, xx.x) |
| | Oninica | Min, Max | XX.X, XX.X | XX.X, XX.X |
| | | Min, Max<br>Mean ± SD | $XX.X \pm XX.X [XX.X, XX.X]$ | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x] |
| | Opinion Seg 3 | Min, Max<br>Mean ± SD<br>N | xx.x ± xx.x [xx.x, xx.x]<br>xx | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx |
| | | Min, Max Mean ± SD N Mean ± SD | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x] |
| | | Min, Max<br>Mean ± SD<br>N | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx |
| | | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max | xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x) | xx.x, xx.x<br>xx.x ± xx.x [xx.x, xx.x]<br>xx<br>xx.x ± xx.x [xx.x, xx.x]<br>xx.x (xx.x, xx.x) |
| | Seg 3 | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max | XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X)<br>XX.X, XX.X | XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX |
| | Seg 3 Opinion | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X] |
| | Seg 3 Opinion | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X]<br>XX.X (XX.X, XX.X)<br>XX.X, XX.X<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X]<br>XX<br>XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 Opinion | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X (XX.X, XX.X) | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX X | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 Opinion | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Mean ± SD | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 Opinion | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 Opinion | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Mean ± SD | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 Opinion Seg 5 | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X, (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X (XX.X, XX.X) XX.X (XX.X, XX.X) XX.X (XX.X, XX.X) |
| | Opinion Seg 4 Opinion Seg 5 Opinion | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X, (XX.X, XX.X) XX.X, ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 Opinion Seg 5 Opinion | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD N Mean ± SD N N Mean ± SD N N Mean ± SD N | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 Opinion Seg 5 Opinion | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 Opinion Seg 5 Opinion | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 Opinion Seg 5 Opinion Seg 6 | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD Median (P25, P75) Min, Max Mean ± SD Median (P25, P75) Min, Max | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 Opinion Seg 5 Opinion Seg 6 | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD Median (P25, P75) Min, Max Mean ± SD Median (P25, P75) Mean ± SD Median (P25, P75) | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] |
| | Opinion Seg 4 Opinion Seg 5 Opinion Seg 6 Opinion Q1/2/3/4/5/6 | Min, Max Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Median (P25, P75) Min, Max Mean ± SD N Mean ± SD N Mean ± SD Median (P25, P75) Min, Max Mean ± SD Median (P25, P75) Min, Max Mean ± SD Median (P25, P75) Min, Max | XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] | XX.X, XX.X XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X (XX.X, XX.X) XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] XX.X ± XX.X [XX.X, XX.X] |

v.1.0; 09-Oct-2020 

### 14.4 Safety Data

# **Table 14.4.1 Immunogenicity**

| Immunoge | enicity | n = xx |
|-----------|--------------|-------------------------|
| V1a (D0) | N | XX |
| | Negative | xx (xx.x%) [xx.x, xx.x] |
| | Positive | xx (xx.x%) [xx.x, xx.x] |
| | Missing Data | XX |
| V3a (D8) | N | XX |
| | Negative | xx (xx.x%) [xx.x, xx.x] |
| | Positive | xx (xx.x%) [xx.x, xx.x] |
| | Missing Data | XX |
| V4a (D29) | N | XX |
| | Negative | xx (xx.x%) [xx.x, xx.x] |
| | Positive | xx (xx.x%) [xx.x, xx.x] |
| | Missing Data | XX |
| V5a (D57) | N | XX |
| | Negative | xx (xx.x%) [xx.x, xx.x] |
| | Positive | xx (xx.x%) [xx.x, xx.x] |
| | Missing Data | XX |
| V6a (D85) | N | XX |
| | Negative | xx (xx.x%) [xx.x, xx.x] |
| | Positive | xx (xx.x%) [xx.x, xx.x] |
| | Missing Data | XX |

95% CI [xx.x, xx.x]

v.1.0; 09-Oct-2020 

**Table 14.4.2 AE Profile Overview – Part B** 

| | | Active (n = xx) | Control<br>(n = xx) | All (n = xx) |
|---|---|---|---|---|
| Participants with any TEAE <sup>a</sup> | Participants | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] |
| | Events | xxx | xxx | xxx |
| Participants with any TRAE <sup>b</sup> | Participants | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] |
| | Events | xxx | xxx | xxx |
| Participants with any SAE <sup>c</sup> | Participants | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] |
| | Events | xxx | xxx | xxx |
| Participants with any TRSAEd | Participants | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] | xx (xx.x%) [xx.x, xx.x] |
| , | Events | XXX | XXX | XXX |

95% CI [xx.x, xx.x]. aTEAE= Treatment-Emergent Adverse Events. bTRAE= Treatment-Related Adverse Events.

Table 14.4.3 Treatment-Emergent AEs Sorted by SOC – Part B

| | | Active<br>(n = xx) | | Control<br>(n = xx) | | All<br>(n = xx) | |
|---|---|---|---|---|---|---|---|
| SOC | PT | Participants | Events | Participants | Events | Participants | Events |
| Any TEAE | | xx (xx.x%) [ xx.x, xx.x] | xx | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| XXXXXXX | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |

95% CI [xx.x, xx.x].

**Table 14.4.4 Treatment-Related AEs Sorted by SOC – Part B** 

| | | Active (n = xx) | | Control<br>(n = xx) | | All<br>(n = xx) | |
|---|---|---|---|---|---|---|---|
| SOC | PT | Participants | Events | Participants | Events | Participants | Events |
| Any TEAE | | xx (xx.x%) [ xx.x, xx.x] | xx | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| XXXXXXX | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |

95% CI [xx.x, xx.x].

v.1.0; 09-Oct-2020 

<sup>°</sup>SAE= Serious Adverse Events. dTRSAE= Treatment-Related Serious Adverse Events.

Table 14.4.5 Treatment-Emergent SAEs Sorted by SOC – Part B

| | | Active<br>(n = xx) | | Control<br>(n = xx) | | All<br>(n = xx) | |
|---|---|---|---|---|---|---|---|
| SOC | PT | Participants | Events | Participants | Events | Participants | Events |
| Any TESAE | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| XXXXXXX | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |

95% CI [xx.x, xx.x].

Table 14.4.6 Treatment-Related SAEs Sorted by SOC – Part B

| | | Active<br>(n = xx) | | Control<br>(n = xx) | | All<br>(n = xx) | |
|---|---|---|---|---|---|---|---|
| SOC | PT | Participants | Events | Participants | Events | Participants | Events |
| Any TRSAE | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | xx | xx (xx.x%) [ xx.x, xx.x] | XX |
| XXXXXX | | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | xx | xx (xx.x%) [ xx.x, xx.x] | XX |
| | XXXXXX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX | xx (xx.x%) [ xx.x, xx.x] | XX |

95% CI [xx.x, xx.x].

v.1.0; 09-Oct-2020 